CLINICAL TRIAL: NCT02501668
Title: The Prevalence of Lung Cancer in Patients With Interstitial Lung Disease
Status: Completed | Type: Observational
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Won-Il Choi, Assoicate Professor, Keimyung University Dongsan Medical Center
Other Study IDs: 2015-05-005
Record Dates: First submitted 2015-07-11; First posted 2015-07-17 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-07

CONDITIONS: Lung Diseases, Interstitial; Lung Cancer
MeSH Terms: conditions — Lung Diseases, Interstitial; Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (11):
- Lung cancer in population: Lung cancer cases in sample population (670,258 cases)
- COPD in population: COPD cases (670,258 cases)
- COPD with lung cancer: Lung cancer in COPD
- ILD without IPF: Interstitial lung disease (ILD) cases without idiopathic pulmonary fibrosis (IPF)
- ILD with lung cancer: Lung cancer cases in ILD
- Idiopathic pulmonary fibrosis: Idiopathic pulmonary fibrosis cases
- IPF with lung cancer: Lung cancer cases in IPF patients
- Connective tissue disorder with ILD: CTD with ILD cases
- CTD ILD with lung cancer: Lung cancer cases in CTD with ILD
- CTD without ILD: CTD with ILD cases in sample population
- CTD without ILD with lung cancer: Lung cancer in CTD without ILD

SUMMARY:
The investigators will evaluate the prevalence of lung cancer associated with interstitial lung disease (ILD) and idiopathic pulmonary fibrosis (IPF) utilizing the Korean Health Insurance Review and Assessment Service (HIRA) database, spanning the period from January 2011 to December 2011. The database (HIRA-NPS-2011-0001) was based on random sampling of outpatients from whole population. Patients with ILDs, IPF, connective tissue disorder (CTD), and COPD were identified based on the International Classification of Disease-10 (ICD-10) diagnostic codes.

DETAILED DESCRIPTION:
The epidemiology of lung cancer related to interstitial lung disease (ILD) with or without with connective tissue disease (CTD) as well as idiopathic pulmonary fibrosis (IPF) has not been well established yet. Interstitial lung disease has a potential to develop lung cancer in the name of scar cancer. The investigators aimed to explore prevalence of lung cancer in patients with ILD with or without CTD and IPF in comparison with chronic obstructive pulmonary disorder (COPD).

The investigators will evaluate the prevalence of lung cancer associated with ILD and IPF utilizing the Korean Health Insurance Review and Assessment Service (HIRA) database, spanning the period from January 2011 to December 2011. The database (HIRA-NPS-2011-0001) was based on random sampling of outpatients from whole population. The sample cases are total 1,375,842. Among them 670,258 cases (age > 40) were evaluated. Patients with ILDs, IPF, CTD, and COPD will be identified based on the International Classification of Disease-10 (ICD-10) diagnostic codes.

ELIGIBILITY:
Inclusion Criteria:

* equal to above 40 years old

Exclusion Criteria:

* none

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a retrospective cohort study based on data collected from the HIRA national database. HIRA is a government-affiliated organization that builds an accurate claims review and is a quality assessment system for the National Health Insurance (NHI). The NHI is the only public medical insurance system operated by the Ministry of Health and Welfare in Korea.
  Korean Health Insurance Review and Assessment Service (HIRA) provided sample database, spanning the period from January 2011 to December 2011. The database (HIRA-NPS-2011-0001) was based on random sampling of outpatients from whole population. The sample cases are total 1,375,842. Among them 670,258 cases (age > 40) were evaluated.
Sampling Method: Probability Sample
Enrollment: 1375842 (Actual)
Dates: Start 2015-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Lung cancer prevalence | Up to 12 months
  Lung cancer prevalence in different groups

CONTACTS AND LOCATIONS:
Overall Officials: Won-Il Choi, MD, Principal Investigator — Keimyung Unversity Dongsan Medical Center